CLINICAL TRIAL: NCT02848521
Title: A Prospective, Non-interventional Study Measuring Quality of Life, Treatment Preference and Treatment Satisfaction of Autosomal Dominant Polycystic Kidney Disease Patients in Europe
Brief Title: A Study Measuring Quality of Life, Treatment Preference and Satisfaction of ADPKD Patients in Europe
Acronym: ACQUIRE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-303-00096
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2018-09

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD; CKD; Rapid progressor; quality of life; DCE
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, non-interventional study (NIS) measuring health-related quality of life (HRQoL), treatment satisfaction, and other patient-reported outcomes (PROs) of ADPKD patients in Europe.

DETAILED DESCRIPTION:
This is a prospective, non-interventional study (NIS) measuring HRQoL, treatment satisfaction, and other PROs of ADPKD patients in Europe. The study aims to enrol at least 486 patients. Data will be prospectively collected at clinics, from medical notes and via PRO measures for each patient at Baseline, Month 1, Month 3 and subsequently at 3 month intervals up to and including the final assessment (18 months maximum follow-up time). No visits with the patients' treating physician will be imposed by the protocol. Any clinical visits will occur as per normal clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged ≥ 18 years.
* Patient has a diagnosis of ADPKD between CKD Stages 1-3, and is deemed by their treating physician to likely have rapidly progressing disease.
* Patient has a life expectancy greater than 18 months at time of enrolment.
* Patient is able and willing to give informed consent, if required according to local regulations.
* Patient is fluent in local language.

Exclusion Criteria:

* Patient is currently participating in, or has in the last 12 months participated in an interventional clinical trial.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient.
* Inability of the patient to complete PROs remotely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients with ADPKD in CKD Stages 1 -3, with evidence of rapidly progressing disease according to the investigator. Investigator must be ADPKD experts qualified by experience and ability to perform the study and be working at an ADPKD reference centre.
Sampling Method: Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Mean rate of change (%) in Physical Health Composite Scale (PCS) scores of the 12-Item Short Form Survey (SF-12) | From Baseline to end of study (maximum of 18 months)
  Mean rate of change (%) in Physical Health Composite Scale (PCS) scores of the SF-12 from baseline to end of study, in the overall sample and per chronic kidney disease (CKD) stage.

SECONDARY OUTCOMES:
Mean rate of change (%) in Mental Health Composite Scale (MCS) scores of the SF-12 | From Baseline to end of study (maximum of 18 months)
  Mean rate of change (%) in Mental Health Composite Scale (MCS) scores of the SF-12 from baseline to end of study, in the overall sample and per CKD stage.
Mean ADPKD-IS score changes | From Baseline to end of study (maximum of 18 months)
  Mean ADPKD-IS scores changes from baseline to end of study, in the overall sample and per CKD stage (physical, emotional and fatigue domain scores will be reported and analysed).
Mean Treatment Satisfaction Questionnaire for Medication (TSQM-9) score changes | From Baseline to end of study (maximum of 18 months)
  Mean TSQM-9 score changes from baseline to end of study, in the overall sample and per CKD stage (effectiveness, convenience and global satisfaction domain scores will be reported and analysed).
Mean ADPKD-Urinary Impact Scale (UIS) score changes | From Baseline to end of study (maximum of 18 months)
  Mean ADPKD-UIS score changes from baseline to end of study, in the overall sample and per CKD stage (frequency, urgency and nocturia domain scores will be reported and analysed).
Description of real-world ADPKD treatment patterns (number of subjects taking different treatments) | From Baseline to end of study (maximum of 18 months)
Description of real-world ADPKD treatment patterns (percentage of subjects taking different treatments) | From Baseline to end of study (maximum of 18 months)

OTHER OUTCOMES:
Mean ADPKD-Pain and Discomfort Scale(PDS) score change from baseline to end of study (exploratory) | From Baseline to end of study (maximum of 18 months)
  Mean ADPKD-PDS score change from baseline to end of study, in the overall sample and per CKD stage (dull kidney pain, sharp kidney pain and fullness/discomfort domain scores will be reported and analysed)
Overall odds ratio of discrete-choice experiment (DCE) for patient preference to the addition of a disease modifying treatment versus no change to local Standard of Care (SoC) | At baseline and at the end of the study (18 months)
  A descriptive of discrete-choice experiment (DCE) will be presented at baseline and at 18 months. Data from the DCE survey will be analysed using a conditional logit model. This explores the impact of each attribute (independent variable) on the patients' choice (dependent variable). Overall odds ratio of DCE for preference to the addition of a disease modifying treatment versus no change to local SoC will be displayed. The relationship between attributes of treatment and overall treatment preference as captured in DCE and relationship between stated DCE attribute preferences and persistence to ADPKD treatments will also be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (26):
- Austria (2):
  - AKH Wien, Vienna
  - LKH Villach, Villach
- Belgium (4):
  - UCL Brussels, Brussels
  - UZ Brussels, Brussels
  - UZ Leuven/Gasthuisberg KUL, Leuven
  - CHU Liège - Domaine Universitaire du Sart Tilman, Liège
- France (5):
  - Clinique La Louviere, Lille
  - CHU Nimes - Hôpital CAREMEAU, Nîmes
  - Hopital Tenon, Paris
  - Necker Hospital, Paris
  - CHU TOURS - Hôpital Bretonneau, Tours
- Germany (3):
  - Charite Berlin, Berlin
  - Universitätsmedizin Göttingen, Göttingen
  - University Medical Center Schleswig-Holstein, Lübeck
- Spain (4):
  - Fundación Puigvert, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de Getafe, Getafe
- Switzerland (2):
  - University Hospital of Geneve, Geneva
  - University Hospital of Zurich, Zurich
- United Kingdom (6):
  - Edinburgh Royal Infirmary, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Aintree University Hospital, Liverpool
  - Royal Free Hospital, London
  - Royal London Hospital, London
  - Freeman Hospital, Newcastle

REFERENCES:
- [Derived] Joly D, Quinn J, Mokiou S, O'Reilly K, Sanchez-Covisa J, Wang-Silvanto J, Doll H. Rationale and study protocol of ACQUIRE, a prospective, observational study measuring quality of life, treatment preference and treatment satisfaction of autosomal dominant polycystic kidney disease (ADPKD) patients in Europe. BMC Nephrol. 2020 Jul 24;21(1):298. doi: 10.1186/s12882-020-01927-1. PMID 32709218